CLINICAL TRIAL: NCT06222762
Title: Effect of a Personalized Follow-up in Adapted Physical Activities on the Long-term Benefits of Rehabilitation in Subjects With Chronic Heart Failure.
Brief Title: Effect of Personalized Follow-up in Adapted Physical Activities in Subjects With Chronic Heart Failure.
Acronym: BougeTonCoeur
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC23.0022 - BOUGE TON COEUR
Record Dates: First submitted 2023-10-26; First posted 2024-01-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial of superiority in parallel arms. Randomised parallel group trial divided into groups according to a ratio (1:1) comparing the follow-up and personalised support after a cardiac rehabilitation programme (experimental group) versus a control group receiving only the usual care, i.e. without follow-up by a sports-health professional (control group), in patients with heart failure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Commun practice (No Intervention): Patient in the control arm will not beneficiate from a follow-up in adapted physical activities (commun practice)
- Follow-up in adapted physical activities (Experimental): Patient in the control arm will beneficiate from a follow-up in adapted physical activities
  Interventions: Other: Experimental arm

INTERVENTIONS:
Other: Experimental arm — Personalized follow-up in adapted physical activities
  Arms: Follow-up in adapted physical activities

SUMMARY:
France has one million people with heart failure (HF). Exercise intolerance, characterised by dyspnoea, is the main clinical symptom in HF patients and a key determinant of reduced quality of life. In addition to drug and surgical treatments, cardiac rehabilitation programmes have shown benefits in heart failure patients. Lasting at least 3 weeks, these programmes improve physical abilities, quality of life and reduce the risk of hospitalisation for heart failure patients.

To date, the real challenge is no longer to prove the benefits of cardiac rehabilitation, but to find solutions to maintain its long-term effects. The transition between the end of the supervised programmes in the centre and the return home is a difficult phase for the majority of patients who do not continue regular physical activity and thus quickly lose the benefits of the programme.

To help maintain the benefits of cardiac rehabilitation, some centres offer patients programmes to continue physical activity during phase III. Although these options are often beneficial in the first few months after the end of rehabilitation compared to control groups, the long-term results are mixed. These results imply that one of these maintenance options may not be suitable for all patients. It is therefore important to propose a personalised post-rehabilitation follow-up involving the patient in the choice of physical activities to optimise the maintenance of long-term benefits.

We hypothesise that patients who receive personalised support from a sport and health professional following rehabilitation maintain long-term benefits compared to a control group who do not receive this support.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable heart failure with NYHA stage I, II or III
* Participation in a cardiac rehabilitation programme
* Patient agreement
* Patient of legal age
* Patient affiliated to the Social Security

Exclusion Criteria:

* Patient refusal
* Minor patients
* Subjects under guardianship or curatorship
* Subjects over 80 years of age at the time of inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2027-09-13 (Estimated); Study Completion 2027-09-13 (Estimated)

PRIMARY OUTCOMES:
To compare the evolution of the level of physical activity 12 months after a cardiac rehabilitation programme between patients benefiting from personalised support at the end of the rehabilitation and a control group benefiting from the usual management. | 12 months
  The primary endpoint will be the difference in mean daily steps measured by accelerometry (over 7 days) at the start of the rehabilitation course (Visit 1) and after 12 months of personalised follow-up (Visit 4).

SECONDARY OUTCOMES:
To compare between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme of time spent in each level of activity : | 12 months
  Levels of activity :
  * Sedentary time (min/day)
  * Time spent in activity with light intensity (min/day)
  * Time spent in activity with moderate intensity (min/day)
  * Time spent in activity with vigorous intensity (min/day)
To compare physical capacities measured using the 6-minute walk test between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  The 6-minute walk test: total walked distance (in metres) The test will be performed twice, the best performance will be kept as reference value.
To compare physical capacities measured using the endurance test between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  The endurance test: endurance time (in seconds) During this test, the patient will be asked to walk at a constant speed (mean speed measured at the 6 minute walking test). If the patient can walk at the requested speed for more than 10 minutes, a second test is performed. The imposed speed is increased by 10% for this second test.
To compare physical capacities measured using the chair getting-up test between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  the total number of time when the patient gets up and sit down on a chair during 1 minute is recorded
To compare physical capacities measured using the hand-grip test between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  The hand-grip test: maximal force (in kg for both hands). the patient will use a dynamometer Hand-grip. The test will be performed 3 times per visit. The force (in Newton) is recorded, the best performance is kept as the reference value
To compare physical capacities measured using the incremental ergocycle test between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  The incremental ergocycle test: maximal power (watts) and VO2 (mL.min.kg-1) The test is performed on a ergocycle.
To compare the evolution of dyspnea scores 12 months after a cardiac rehabilitation programme between the experimental group and the control group | 12 months
  Dyspnea-12 questionnaire dyspnea scores DYSPNEA 12 : The DYSPNEA 12 comprised of 12 different breathlessness descriptors with each scored on a four-item scale (none-0, mild-1, moderate2, severe-3). Item scores are summed (D-12 Total) and can be divided into sub-scores reflecting Physical and Affective domains.
To compare the psychological dimensions (motivation) between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  EMAPS questionnaire EMAPS : The questionnaire includes 18 items. The EMAPS is used to evaluate the motivation to practice physical activities. The answer to questions goes from 1 to 7 with 1 (does not match at all) and 7 (matches very strongly).
To compare the psychological dimensions (anxiety/depression) between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  HAD questionnaire HAD : The questionnaire includes 7 items for depression and 7 items for anxiety. Each item had been answered by the patient on a four point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and for depression. A score of 0 to 7 for either subscale could be regarded as being in the normal range, a score of 11 or higher indicating probable presence ('caseness') of the mood disorder and a score of 8 to 10 being just suggestive of the presence of the respective state.
To compare the psychological dimensions (quality of life) between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  SF-36 : The Short Form 36 (SF36) is used to evaluate the quality of life. The SF36 scale includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue)
To compare the psychological dimensions (quality of life) between the experimental group and the control group, the evolution 12 months after a cardiac rehabilitation programme | 12 months
  EQ5D5L : The questionnaire includes 5 items mobility, personal care, usual activities, pain/discomfort and anxiety/depression.
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the physiological adaptations during endurance test | 12 months
  Comparison of physiological adaptations assessed in the endurance test
  - Ventilatory parameters (minute ventilation, respiratory rate and tidal volume)
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the physiological adaptations during endurance test | 12 months
  Comparison of physiological adaptations assessed in the endurance test
  - Gas exchange (VO2, VCO2)
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the physiological adaptations during endurance test | 12 months
  Comparison of physiological adaptations assessed in the endurance test
  - Cardio-ventilatory parameters (heart rate in beat/min and electrocardiogram (ECG))
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the physiological adaptations during endurance test | 12 months
  comparison of physiological adaptations assessed in the incremental test:
  - Ventilatory parameters (minute ventilation, respiratory rate and tidal volume)
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the physiological adaptations during endurance test | 12 months
  comparison of physiological adaptations assessed in the incremental test:
  - Gas exchange parameters (VO2, VCO2)
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the physiological adaptations during endurance test | 12 months
  comparison of physiological adaptations assessed in the incremental test:
  - Cardiovascular parameters (heart rate in beat/min, electrocardiogram (ECG), systolic and diastolic pression (mmHg)
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the endothelial dysfunction : microcirculation | 12 months
  - Analyse of skin circulation (laser doppler) with post-occlusive reactive hyperemia et hyperthermia
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the endothelial dysfunction : macrocirculation | 12 months
  - Analyse by flow-mediated dilatation (FMD) by echography
To compare, between groups, the evolution 12 months after a cardiac rehabilitation programme of the endothelial dysfunction : blood markers | 12 months
  - Analyses of several blood markers related to endothelial dysfunction, inflammation and/or heart failure : IL-6 ; IL-10; VEGF-A; Ang-1; Ang-2; IL-1β; TNF-α; MCP-1; IL-8; EGF; E-selectine; I-CAM 1; PECAM-1; VCAM-1; tPA; CRP; VWF; NT-pro-BNP; ET-1

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Mansourati, MD, PhD, Principal Investigator — Brest Universty Hospital
Locations (2):
- France (2):
  - Fondation ILDYS, Brest
  - CHU de Brest, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement